CLINICAL TRIAL: NCT05178433
Title: Randomized Controlled Study of Skin Care Strategies for Neonatal Jaundice Phototherapy to Prevent Atopic Dermatitis in Moderate and Severe Infants
Brief Title: Skin Care Strategies for Neonatal Jaundice Phototherapy to Prevent Atopic Dermatitis in Moderate and Severe Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ShanghaiFMIH-KS21259
Record Dates: First submitted 2021-11-22; First posted 2022-01-05 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Neonatal Jaundice; Atopic Dermatitis
MeSH Terms: conditions — Jaundice, Neonatal; Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Use baby moisturizers in addition to basic skin care and protection during phototherapy.
  Interventions: Combination Product: Use baby moisturizers by NeoChine
- control group (No Intervention): Only basic skin care and protection during phototherapy.

INTERVENTIONS:
Combination Product: Use baby moisturizers by NeoChine — During continuous phototherapy, use skin basic care and protection in combination with baby moisturizing products, use the whole body twice a day, and the amount of each time is not less than 5 grams.
  Arms: Experimental group

SUMMARY:
Atopic Dermatitis (AD) is a common chronic, recurrent, and inflammatory skin disease in children. The incidence of moderate to severe AD in infants aged 1-12 months in our country is as high as 25.41%, which is related to subsequent allergic diseases and affects Children's emotions and growth. There are limited drugs that can be used for infant AD. The current guidelines recommend early use of functional skin care products to prevent and treat AD by repairing the skin barrier, moisturizing, and anti-inflammatory. Neonatal jaundice is one of the most common neonatal diseases. 20% of children with jaundice need phototherapy. It is a simple and effective method for jaundice. Studies have found that phototherapy can convert Th2 to Th1, leading to an imbalance of pro-inflammatory and anti-inflammatory, which induces allergies. We speculate that it is of great value to take protective measures such as skin moisturizing during phototherapy for jaundice in children at high risk of allergies. This project intends to take the lead in conducting a randomized controlled study on the use of baby moisturizing products during neonatal phototherapy. Through evaluation projects such as skin microecology analysis, serum allergy indicators and AD clinical manifestations, it is verified that the use of functional skin care products in phototherapy of newborns with high allergies can delay and reduce the severity of AD in infants.

DETAILED DESCRIPTION:
Atopic Dermatitis (AD) is a common chronic, recurrent, and inflammatory skin disease. The onset before 1 year old accounts for about 50% of all patients. The main manifestations are dry skin, chronic eczema-like dermatitis and severe itching. The incidence of AD in infants worldwide is as high as 30%. In our country, the prevalence of AD among infants aged 1-12 months is 30.48%, of which 23.97% are moderate and 1.44% are severe. Infant AD is mostly related to non-IgE-mediated food allergies. The prevalence rate of food allergy in children with moderate to severe AD under 2 years of age in our country is 49.7% confirmed by food provocation test, which seriously affects the nutritional intake and growth and development of children. Cause psychological and economic burdens on children and their families. At present, AD is considered to be a multifactorial disease, involving genetic susceptibility, immune disorders, microbial flora imbalance, environmental factors, and skin barrier function defects. Different from adults, the immune system of infants and young children is not yet mature. AD, allergic asthma and allergic rhinitis are known as the triad of children's atopic. Among them, AD is the earliest age of onset. It may be the first step in the process of allergic diseases. It is unique The pathogenesis related research is relatively limited, and there are only a handful of drugs approved for infantile AD. Therefore, the prevention of moderate to severe infantile AD should be more important than treatment.

Neonatal jaundice is one of the most common neonatal disorders. The incidence of full-term infants within one week of birth is 60%, and premature infants are as high as 80%. Among them, in order to prevent and treat bilirubin encephalopathy, children with severe neonatal hyper-indirect bilirubinemia need to receive phototherapy. The most commonly used blue light therapy in clinical practice is a simple, effective and relatively safe measure to reduce jaundice. About 20% of children with jaundice receive phototherapy. Bilirubin is an antioxidant that can neutralize free radicals produced in the body after birth. The imbalance of the body's oxidation-antioxidation mechanism may cause allergic diseases. Studies have focused on the occurrence and development of neonatal jaundice and allergic diseases. At the same time, blue light therapy is suitable for moderate to severe neonatal hyperbilirubinemia, which can cause the rapid conversion of Th2 to Th1, thereby increasing the pro-inflammatory factor tumor necrosis factor-α (TNF-α), interleukin-8 (IL- 8) and IL-1β, and reduce IL-6 and other anti-inflammatory factors, thereby exacerbating the inflammatory process and allergic diseases. Some recent studies suggest that children with neonatal jaundice are more likely to develop allergic diseases than those without jaundice, and the incidence is 14.1% higher; early-onset neonatal jaundice is positively correlated with blue light therapy in the occurrence and development of allergic diseases. Therefore, it is of great clinical significance to take protective measures to reduce or delay the occurrence of moderate to severe AD in infants and young children when blue light treatment is required for jaundice in children at high risk of allergies.

At the same time, common adverse reactions of neonatal phototherapy include skin rash, fever, diarrhea, etc., and long-term damage to the DNA of skin cells. In order to avoid damaging the health of infants, it is indeed necessary to further standardize and rationalize phototherapy. Infant functional skin care products have the functions of repairing the skin barrier, moisturizing, and anti-inflammatory, and are important basic treatment methods for children with AD. Studies have pointed out that topical moisturizers should be used as early as possible in the neonatal period to reduce and postpone the occurrence of AD. At present, only sensitive parts such as eyes, external genitalia, or vulva should be covered during phototherapy of newborns. There is no research published on skin protection measures during phototherapy.

In summary, neonatal jaundice and phototherapy due to jaundice are very likely to be related to the occurrence and development of infantile AD, and AD is the earliest allergic disease. The relevant clinical guidelines point out that the early standardized use of infant moisturizing products can reduce the occurrence of moderate to severe AD. . Therefore, this project intends to take the lead in conducting research on skin care for newborns at high risk of allergies who need phototherapy. This study is a randomized controlled study. It intends to randomly provide baby moisturizing product care for allergic high-risk newborns who need phototherapy, and verify skin moisturizing during phototherapy of allergic high-risk newborns through evaluation items such as skin microecology analysis, serum allergy indicators, and AD clinical manifestations. It is an effective measure to delay and reduce the severity of AD in infancy.

ELIGIBILITY:
Inclusion Criteria:

1. Full-term newborns who were admitted to the hospital with phototherapy were treated with "neonatal hyperbilirubinemia".
2. Ask about a positive family history of allergic diseases, that is, the parents and siblings are atopic constitutions, including allergic asthma, allergic rhinitis, allergic conjunctivitis and (or) history of AD, as well as a significant increase in IgE.
3. The guardian voluntarily followed the doctor's guidance for treatment and follow-up during the entire study period, and signed an informed consent form.
4. Exclude severe heart, brain, lung, kidney disease and fatal congenital malformations.

Exclusion Criteria:

1. Those who do not meet the selection criteria or meet the exclusion criteria after review.
2. After enrollment, due to the disease, the jaundice gradually worsened to reach the indications for transfusion therapy.
3. Other skin diseases other than infant AD were diagnosed during the follow-up period.
4. Guardians voluntarily withdraw from the study.

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The effect of using external moisturizing products for infants and young children on the occurrence of moderate to severe AD within 6 months of age. | up to 6 months
  The Chinese children's AD diagnostic criteria, combined with the SCORAD score, were used to find the diagnosis and severity of AD in newborns up to 6 months of age, and to compared whether skin care interventions during phototherapy have an effect on delaying and lowering AD.

SECONDARY OUTCOMES:
The effect of external moisturizing products on phototherapy | up to 6 months
  The amount of water loss in the epidermis and the water content in the stratum corneum was obtained by measuring the water loss of the skin, compare changes before and after phototherapy, and compare with infants who use baby moisturizing products during phototherapy to see if there is a difference in skin barrier function between the two groups of children.
The effect of jaundice phototherapy on the skin microecology of allergic high-risk infants | up to 6 months
  During the admission and discharge of phototherapy, the skin microbiota metagenomic sequencing was performed by taking skin swabs from the children's forehead.
The effect of phototherapy on the level of neonatal inflammatory factors | up to 6 months
  Detection of serum tumor necrosis factor-α (TNF-α), interleukin-2 (IL-2), IL-6, IL-8 and IL-10 levels

CONTACTS AND LOCATIONS:
Overall Officials: Li Jing, Study Director — Shanghai First Maternity and Infant Health Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langan SM, Irvine AD, Weidinger S. Atopic dermatitis. Lancet. 2020 Aug 1;396(10247):345-360. doi: 10.1016/S0140-6736(20)31286-1. PMID 32738956
- [Background] Drucker AM, Wang AR, Li WQ, Sevetson E, Block JK, Qureshi AA. The Burden of Atopic Dermatitis: Summary of a Report for the National Eczema Association. J Invest Dermatol. 2017 Jan;137(1):26-30. doi: 10.1016/j.jid.2016.07.012. Epub 2016 Sep 8. PMID 27616422
- [Background] Guo Y, Zhang H, Liu Q, Wei F, Tang J, Li P, Han X, Zou X, Xu G, Xu Z, Zong W, Ran Q, Xiao F, Mu Z, Mao X, Ran N, Cheng R, Li M, Li C, Luo Y, Meng C, Zhang X, Xu H, Li J, Tang P, Xiang J, Shen C, Niu H, Li H, Shen J, Ni C, Zhang J, Wang H, Ma L, Bieber T, Yao Z. Phenotypic analysis of atopic dermatitis in children aged 1-12 months: elaboration of novel diagnostic criteria for infants in China and estimation of prevalence. J Eur Acad Dermatol Venereol. 2019 Aug;33(8):1569-1576. doi: 10.1111/jdv.15618. Epub 2019 May 17. PMID 30989708
- [Background] Yang H, Xiao YZ, Luo XY, Tan Q, Wang H. Diagnostic accuracy of atopy patch tests for food allergy in children with atopic dermatitis aged less than two years. Allergol Immunopathol (Madr). 2014 Jan-Feb;42(1):22-8. doi: 10.1016/j.aller.2012.10.007. Epub 2012 Dec 17. PMID 23253686
- [Background] Low DW, Jamil A, Md Nor N, Kader Ibrahim SB, Poh BK. Food restriction, nutrition status, and growth in toddlers with atopic dermatitis. Pediatr Dermatol. 2020 Jan;37(1):69-77. doi: 10.1111/pde.14004. Epub 2019 Oct 30. PMID 31667896
- [Background] Vakharia PP, Silverberg JI. New and emerging therapies for paediatric atopic dermatitis. Lancet Child Adolesc Health. 2019 May;3(5):343-353. doi: 10.1016/S2352-4642(19)30030-6. Epub 2019 Mar 20. PMID 30904349
- [Background] Nadeem A, Masood A, Siddiqui N. Oxidant--antioxidant imbalance in asthma: scientific evidence, epidemiological data and possible therapeutic options. Ther Adv Respir Dis. 2008 Aug;2(4):215-35. doi: 10.1177/1753465808094971. PMID 19124374
- [Background] Das RR, Naik SS. Neonatal hyperbilirubinemia and childhood allergic diseases: a systematic review. Pediatr Allergy Immunol. 2015 Feb;26(1):2-11. doi: 10.1111/pai.12281. Epub 2014 Oct 13. PMID 25229699
- [Background] Procianoy RS, Silveira RC, Fonseca LT, Heidemann LA, Neto EC. The influence of phototherapy on serum cytokine concentrations in newborn infants. Am J Perinatol. 2010 May;27(5):375-9. doi: 10.1055/s-0029-1243311. Epub 2009 Dec 11. PMID 20013604
- [Background] Beken S, Aydin B, Zencirogglu A, Dilli D, Ozkan E, Dursun A, Okumus N. The effects of phototherapy on eosinophil and eosinophilic cationic protein in newborns with hyperbilirubinemia. Fetal Pediatr Pathol. 2014 Jun;33(3):151-6. doi: 10.3109/15513815.2014.883456. Epub 2014 Feb 14. PMID 24527832
- [Background] Safar H, Elsary AY. Neonatal Jaundice: The Other Side of the Coin in the Development of Allergy. Am J Perinatol. 2020 Nov;37(13):1357-1363. doi: 10.1055/s-0039-1693697. Epub 2019 Jul 31. PMID 31365932
- [Background] Wang J, Guo G, Li A, Cai WQ, Wang X. Challenges of phototherapy for neonatal hyperbilirubinemia (Review). Exp Ther Med. 2021 Mar;21(3):231. doi: 10.3892/etm.2021.9662. Epub 2021 Jan 20. PMID 33613704
- [Result] Horimukai K, Morita K, Narita M, Kondo M, Kitazawa H, Nozaki M, Shigematsu Y, Yoshida K, Niizeki H, Motomura K, Sago H, Takimoto T, Inoue E, Kamemura N, Kido H, Hisatsune J, Sugai M, Murota H, Katayama I, Sasaki T, Amagai M, Morita H, Matsuda A, Matsumoto K, Saito H, Ohya Y. Application of moisturizer to neonates prevents development of atopic dermatitis. J Allergy Clin Immunol. 2014 Oct;134(4):824-830.e6. doi: 10.1016/j.jaci.2014.07.060. PMID 25282564
- [Result] Cheng R, Zhang H, Zong W, Tang J, Han X, Zhang L, Zhang X, Gu H, Shu Y, Peng G, Huang L, Liu Q, Gao X, Guo Y, Yao Z. Development and validation of new diagnostic criteria for atopic dermatitis in children of China. J Eur Acad Dermatol Venereol. 2020 Mar;34(3):542-548. doi: 10.1111/jdv.15979. Epub 2019 Oct 31. PMID 31568595